CLINICAL TRIAL: NCT02115139
Title: A Multicenter, Single Arm, Phase 2 Clinical Study on the Combination of Radiation Therapy and Ipilimumab, for the Treatment of Patients With Melanoma and Brain Metastases
Brief Title: GEM STUDY: Radiation And Yervoy in Patients With Melanoma and Brain Metastases
Acronym: GRAY-B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM 1202; 2013-001132-22 (EudraCT Number)
Record Dates: First submitted 2014-04-10; First posted 2014-04-15 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Melanoma; Brain Metastases
Keywords: melanoma; brain; metastases; Patients with melanoma and brain metastases
MeSH Terms: conditions — Melanoma; Brain Neoplasms; Neoplasm Metastasis | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipilimumab (Experimental): Ipilimumab 3mg/Kg iv q 3 weeks for 4 cycles Whole-brain radiotherapy (WBRT) 30 Gy in 10 fractions (or radiobiological equivalent schedule, after Sponsor approval), starting between Cycle 1 Day 2 and Cycle 2 Day 1
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 3mg/Kg iv q 3 weeks for 4 cycles
  Other Names: Experimental

SUMMARY:
Ipilimumab adds a clinical benefit to radiation therapy in patients with melanoma metastatic to the brain.

Melanoma is the third most common cancer causing brain metastases, after cancers of the lung and breast, which appears to reflect the relative propensity of melanoma to metastasize to the central nervous system (CNS). Brain metastases are responsible for 20 to 54 percent of deaths in patients with melanoma, and among those with documented brain metastases, these lesions contribute to death in up to 95 percent of cases, with an estimated median overall survival ranging between 1.8 and 10.5 months, depending upon other prognostic factors.

Ipilimumab is an anti-Cytotoxic T-Lymphocyte Antigen 4 (anti-CTLA4) monoclonal antibody that has demonstrated a clinically relevant and statistically significant improvement in overall survival, either alone (second line) or in combination with dacarbazine (DTIC) in 1st line.

Ipilimumab has shown activity against brain metastases.

According to the European Medicines Agency (EMA) approved label for Yervoy®, the use of glucocorticoids at baseline (commonly prescribed when brain metastases are diagnosed) should be avoided before the administration of ipilimumab. Data show that the use of even high doses of glucocorticoids for the management of immune-related adverse events do not decrease the efficacy of Yervoy®. There is no documented experience on the efficacy of Yervoy® when given concomitantly with radiation therapy and glucocorticoids.

In experimental models, radiation therapy is synergistic to anti-Cytotoxic T-Lymphocyte Antigen 4 (anti-CTLA4) strategies (abscopal effect).

There are no published results from clinical trials on the interaction between radiation therapy and ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent.
2. Histologic diagnosis of melanoma.
3. First episode of radiological evidence of brain metastases
4. Be over the age of 18 years old
5. Radiation Therapy Oncology Group-recursive partitioning analysis (RTOG-RPA) class 2
6. Karnofsky performance status (PS) more than 70%
7. Barthel Index of Activities of Daily Living more than 10
8. Measurable disease (mWHO criteria).
9. Adequate organ function as determine by the following criteria:

   * White blood count (WBC) more or equal to 2000/ microliter (uL)
   * Absolute neutrophil count (ANC) more than 1.5 x 109/L.
   * Platelet count more than 75 x 109/L.
   * Hemoglobin more than 9 g/dL. If the patient received a red blood count (RBC) transfusion, the required value of hemoglobin should be met at least 1 week after the most recent transfusion.
   * Serum creatinine less or equal to 2.0 x upper limit of normal (ULN).
   * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) less or equal to 2.5 x ULN for patients without liver metastasis, or less or equal to 5 times for liver metastases.
   * Total bilirubin less or equal 2.0 x ULN, (except patients with Gilbert's Syndrome, who must have a total bilirubin less than 3.0 mg/dL)
10. Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 26 weeks after ipilimumab is stopped

Exclusion Criteria:

1. Patients with melanoma and brain metastases with any of the following disease-specific characteristics:

   * Documented evidence of prior progression of melanoma to an ipilimumab-containing regimen (i.e. received at least 2 doses of ipilimumab for either advanced disease or in the adjuvant setting and the disease progressed/relapsed (according to mWHO criteria) within 24 weeks since the first dose of ipilimumab)
   * Prior radiation therapy to the brain
   * Other prior antineoplastic therapies for brain metastases.
   * Patients with cerebral metastases as the only location of the disease, for which local therapy (neurosurgery, radiosurgery) could achieve a disease-free status
   * Patients with a rapid clinical deterioration, or with risk of herniation, or who require unstable ascending dosing of supportive medication in the last week -including anti-convulsivants, steroids and analgesics-, or who require dexamethasone more than 16 mg/d (or other glucocorticoid at an equipotent dose), or with a high lactate dehydrogenase (LDH) more than 2 x ULN.
2. Any other malignancy form which the patient has been disease-free for less than 5 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix, or incidental prostate cancer.
3. Uncontrolled diabetes mellitus (HbA1c more than 9 %)
4. Autoimmune disease other than vitiligo or past thyroiditis under substitutive hormone therapy: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
5. Other chronic intestinal diseases associated with diarrhea.
6. Active infection or other serious illness or medical condition.
7. Known active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
8. Concomitant therapy with any of the following: interleukin-2 (IL-2), interferon, or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids (used for the management of non-cancer related illnesses), either concomitantly or during the last 30 days prior to the beginning of the treatment.
9. Any experimental therapy administered in the past 30 days prior to the beginning of the treatment.
10. Any non-oncology vaccine therapy used for the prevention of infectious diseases (for up to 4 weeks prior to or after any dose of blinded study drug) (see definitions in protocol text)
11. Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness.
12. Any other general, medical or psychological conditions which in the opinion of the investigator will make the administration of ipilimumab hazardous, or that would preclude appropriate informed consent or compliance with the protocol, or obscure the interpretation of eventual adverse events (AEs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-04-04 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: José A López-Martín, MD, Study Chair — Hospital Universitario 12 de Octubre - GEM
Locations (12):
- Spain (12):
  - ICO Badalona, Badalona
  - H. Clinic de Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - H. Insular de Canarias, Las Palmas de Gran Canaria
  - H. U. Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - H. Clínico de Santiago, Santiago de Compostela
  - H.U. Virgen Macarena, Seville
  - H. Virgen de la Salud, Toledo
  - H. General de Valencia, Valencia
  - Instituto Valenciano de Oncología, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 patients were enrolled and fulfilled the inclusion criteria, analyzed for safety.
  During the trial 7 patients discontinued treatment before completion, so the total of patients for efficacy analysis was 51.
Period: Overall Study
Arm/Group | Ipilimumab
Started | 58
Completed | 51
Not Completed | 7
Not completed — Protocol Violation | 1
Not completed — treatment discontinuation | 6

BASELINE CHARACTERISTICS:
Arm/Group | Ipilimumab
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: Years] | 66 [36.8 to 84.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 36
Region of Enrollment [Count of Participants; unit: Participants]
  Spain | 58
Karnofsky performance status (KPS) [Count of Participants; unit: Participants] — Karnofsky performance status (KPS) allows patients to be classified as to their functional impairment. The scale ranges from 0 (death, worst performance) to 100 (complete functional, better performance).
  Participants
    90-100 | 42
    70-80 | 15
    Not evaluable (NE) | 1
Barthel index [Count of Participants; unit: Participants] — Barthel index measures the capacity of the person for the execution of ten basic activities in daily life. The index ranges from 0 (worst performance) to 20 (best performance).
  Participants
    Lower than 15 | 2
    15-20 | 56
BRAF mutational status [Count of Participants; unit: Participants]
  Mutated | 20
  Native | 30
  Not evaluated (NE) | 8
Number of previous treatment lines [Count of Participants; unit: Participants]
  No previous lines | 29
  1 previous line | 20
  2 or more previous lines | 9
Number of brain metastasis [Count of Participants; unit: Participants]
  Single brain lesion | 14
  Multiple brain lesions | 43
  Not especified (NE) | 1
Corticoid use [Count of Participants; unit: Participants]
  Yes | 25
  No | 33
Lactate dehydrogenase (LDH) blood levels [Count of Participants; unit: Participants]
  Levels higher than Upper limit normal (ULN): Yes | 24
  Levels higher than Upper limit normal (ULN): No | 34
  Levels higher than 1.5X Upper limit normal (ULN): Yes | 9
  Levels higher than 1.5X Upper limit normal (ULN): No | 49

OUTCOME MEASURES:

1. Primary Outcome: 1-year Survival Rate
Description: During treatment period, there will be assessments every cycle. After end of treatment every 3 month.
Time Frame: From date of inclusion until the date of first documented date of death from any cause, assessed every 3 weeks during for the first 6 months, then every 3 months. Up to 1 year
Population: Efficacy cohort, all patients that fulfill eligibility and completed the treatment with radiotherapy
Measure: Number (95% Confidence Interval); unit: Percentage of patients alive at 1 year
Arm/Group | Ipilimumab
Number analyzed (Participants) | 51
Percentage of patients alive at 1 year | 31.8 [18.8 to 44.8]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Median time from treatment initiation to progression of disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Within 4 weeks before start treatment, week 12, 17+/-1 and every 9 + / -1 weeks until progression up to 12 months after last patient treatment initiation.
Population: Efficacy population (patients that fulfill eligibility and completed the treatment with radiotherapy)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab
Number analyzed (Participants) | 51
Months | 3.11 [2.23 to 3.98]

3. Secondary Outcome: Intracranial PFS
Description: median, 6-month PFS rate
Time Frame: as for outcome 2
Population: Data were not collected
Arm/Group | Ipilimumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Extracranial PFS
Description: median, 6-month PFS rate
Time Frame: as for outcome 2
Population: Data were not collected
Arm/Group | Ipilimumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: median value for OS estimated by kaplan meier method
Time Frame: From date of inclusion until the date of first documented date of death from any cause, assessed every 3 weeks during for the first 6 months, then every 3 months.
Population: Efficacy population (patients that comply with eligibility and completed radiotherapy treatment)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab
Number analyzed (Participants) | 51
Months | 4.73 [3.59 to 5.87]

6. Secondary Outcome: Response Rate
Description: Measured according to Who response criteria and Immune-related response criteria.
  Response for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: as for outcome 2
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 51
Participants
  modified WHO criteria: Complete Response (CR) | 2
  modified WHO criteria: Partial response (PR) | 3
  modified WHO criteria: Stable disease (SD) | 12
  modified WHO criteria: Progression disease (PD) | 19
  modified WHO criteria: Not evaluable (NE) | 15
  Immun related response criteria (irRC): Complete Response (CR) | 2
  Immun related response criteria (irRC): Partial response (PR) | 3
  Immun related response criteria (irRC): Stable disease (SD) | 12
  Immun related response criteria (irRC): Progression disease (PD) | 17
  Immun related response criteria (irRC): Not evaluable (NE) | 17

7. Secondary Outcome: Adverse Event Rates
Description: Number of patients with at least one treatment-related toxicity, classified by grade.
Time Frame: From date of inclusion until the date of first documented date of death from any cause or end of study, assessed every 3 weeks during for the first 6 months, then every 3 months.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 58
Participants
  Any grade toxicity: Yes | 37
  Any grade toxicity: No | 21
  Grade 3 or higher toxicity: Yes | 11
  Grade 3 or higher toxicity: No | 47

8. Secondary Outcome: Rate of Dose Delays/Reductions and Treatment Exposure.
Description: Treatment feasibility. Number of patients with treatment delays and reductions, categorized as function of the number of events (reductions/delays)
Time Frame: Expected average of 3 weeks during for the first 6 months, then every 3 months.
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 58
Participants
  Ipilimumab delay: None | 43
  Ipilimumab delay: 1 event | 12
  Ipilimumab delay: 2 events | 2
  Ipilimumab delay: 3 events | 1
  Ipilimumab delay: 4 events | 0
  Ipilimumab reductions: None | 50
  Ipilimumab reductions: 1 event | 5
  Ipilimumab reductions: 2 events | 1
  Ipilimumab reductions: 3 events | 1
  Ipilimumab reductions: 4 events | 1

9. Other Pre Specified Outcome: Correlation of Biomarker Expression and PFS.
Description: Translational study. PFS outcome reported by subgroups according to BRAF mutation status
Time Frame: Within 28 days before start treatment, just before the start treatment, then expected average of 3 weeks for the first 12 weeks
Population: efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab
Number analyzed (Participants) | 51
Participants
  BRAF mutated: Progression disease | 5
  BRAF mutated: No progression | 12
  BRAF mutated: Not applicable | 34
  BRAF native: Progression disease | 7
  BRAF native: No progression | 19
  BRAF native: Not applicable | 25

10. Other Pre Specified Outcome: Intrapatient Variation of Quantitative Apparent Diffusion Coefficients of Serial Diffusion-weighted Magnetic Resonance Imaging
Time Frame: Baseline and 4 weeks after WBRT
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Throughout the study period, from inclusion to 30 days after treatment has ended. Approximately 1 year
Arm/Group | Ipilimumab
All-Cause Mortality (participants affected / at risk) | 40/58
Serious Adverse Events (participants affected / at risk) | 33/58
Other Adverse Events (participants affected / at risk) | 57/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=58)
Anemia (Blood and lymphatic system disorders) | 1
Ataxia (Nervous system disorders) | 1
Blood bilirrubin increase (Investigations) | 1
Cognitive disturbance (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Dizziness (Nervous system disorders) | 1
Dysphasia (Nervous system disorders) | 1
Hemianopsia (Eye disorders) | 1
Fever (General disorders) | 2
Gastric Hemorrage (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Candidiasis (Infections and infestations) | 1
Intracranial hemorrage (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 2
Malaise (General disorders) | 4
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Pleural effussion (Respiratory, thoracic and mediastinal disorders) | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Seizures (Nervous system disorders) | 2
Sepsis (Infections and infestations) | 1
somnolence (Nervous system disorders) | 1
Testicular disorder (Reproductive system and breast disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Vomiting (Gastrointestinal disorders) | 2
Hepatotoxicity (Hepatobiliary disorders) | 1
Depression (Psychiatric disorders) | 1
Duodenal perforation (Gastrointestinal disorders) | 1
ALT increased (Investigations) | 1
GPT increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab (N=58)
Alopecia (Skin and subcutaneous tissue disorders) | 9
Anorexia (Metabolism and nutrition disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 14
Dizziness (Nervous system disorders) | 7
Edema (Blood and lymphatic system disorders) | 6
Fatigue (General disorders) | 28
Fever (General disorders) | 7
Headache (Nervous system disorders) | 23
Hyperglycemia (Metabolism and nutrition disorders) | 6
Nausea (Gastrointestinal disorders) | 16
Pruritus (Skin and subcutaneous tissue disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 5
Vomiting (Gastrointestinal disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2013-11-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT02115139/Prot_000.pdf
  • Statistical Analysis Plan (2013-11-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT02115139/SAP_001.pdf